CLINICAL TRIAL: NCT03278665
Title: An Open-label Phase Ib/II, Multi-center Study of 4SC-202 in Combination With Pembrolizumab in Patients With Unresectable Stage III/Metastatic Stage IV Cutaneous Melanoma Primary Refractory/Non-responding to Prior Anti-PD-1 Therapy
Brief Title: 4SC-202 in Combination With Pembrolizumab in Patients Primary Refractory/Non-responding to Prior Anti-PD-1 Therapy
Acronym: SENSITIZE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 4SC AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-202-2-2017
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Malignant Melanoma
Keywords: Cutaneous melanoma
MeSH Terms: conditions — Melanoma | interventions — domatinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SC-202 + Pembrolizumab (Experimental): Single arm study of 4SC-202 in combination with Pembrolizumab
  Interventions: Drug: 4SC-202 in combination with Pembrolizumab

INTERVENTIONS:
Drug: 4SC-202 in combination with Pembrolizumab — 4SC-202 in combination with Pembrolizumab

SUMMARY:
Phase Ib/II open-label, multi-center study with a priming cycle of 4SC-202 to evaluate the safety, tolerability and preliminary efficacy of combination treatment with 4SC-202 and Pembrolizumab. A dose expansion cohort at the Recommended Phase Two Dose (RPTD) will be added.

Adult patients with advanced (unresectable or metastatic) cutaneous melanoma primary refractory or non-responding to anti-PD-1 therapy as most current systemic anti-cancer therapy and for whom no standard therapy is available, will be enrolled. The last administration of anti-PD-1 therapy must have been performed within 6 months prior to screening.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with unresectable stage III or stage IV cutaneous melanoma, as per American Joint Committee on Cancer (AJCC) (Version 8) staging system (must have been histologically confirmed at least once during course of disease). Patients with metastatic tumor of unknown primary site and histology of melanoma are eligible.
* Patients must be primary refractory or non-responding to anti-PD-1 therapy (either as monotherapy or in combination with Ipilimumab)
* Measurable disease by computer tomography (CT) or Magnetic resonance imaging (MRI) per immune-related response evaluation criteria in solid tumors (irRECIST) 1.1 criteria, with longest diameter for non-nodal lesions ≥ 10 mm and ≥ 15 mm in short axis for nodal lesions
* At least one tumor site (either primary site or metastasis) must be accessible for sequential biopsies and patient must consent to the 2 mandatory biopsies. This requirement is not applicable for continuous dosing schedules and may be waived by the sponsor in other individual cases.

Main Exclusion Criteria:

* Patients who achieved a CR or PR, during or after prior anti-PD-1 mono- or anti-CTLA-4/anti-PD-1 combination therapy
* Patients with symptomatic brain metastases/central nervous system (CNS) involvement
* Patients with inadequate organ function
* Therapy with agents known to prolong the QT interval and increase the risk for Torsades de Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | Up to 114 weeks
  Safety and tolerability of the combination of 4SC-202 and Pembrolizumab will be assessed from adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 102 weeks
  The Objective Response Rate (ORR) will be defined as the percentage of patients who have achieved a confirmed response of at least Immune-related Complete Response (irCR) or Immune-related Partial Response (irPR)
Best Overall Response (BOR) | Up to 102 weeks
  The Best Overall Response defined as the best among all confirmed overall responses (irCR is better than irPR is better than irSD)
Disease Control Rate (DCR) | Up to 102 weeks
  The Disease Control Rate (DCR) will be defined as the percentage of patients who have achieved a confirmed response of at least irCR or irPR or a response of irSD
Duration of Response (DOR) | Up to 102 weeks
  Duration of response (DOR) is defined as the time from the first documentation of response to the date of disease progression. Patients who have no documented disease progression at the end of the study or who are lost to follow-up or who receive additional anti-neoplastic therapy after discontinuing 4SC-202 and Pembrolizumab will be censored at the date of their last extent of disease assessment or on the first date of additional therapy, respectively.
Progression Free Survival (PFS) | Up to 102 weeks
  The time from first dosing (C1D1) to date of first observed progression or death from any cause (whichever comes first). Patients who have not progressed while on study and have not died while on study will be censored at the last evaluable assessment date.
Time to Progression (TTP) | Up to 102 weeks
  The time from first dosing (C1D1) to first date of first observed progression. Patients who have not progressed while on study, have not died while on study or experienced a non-disease- related death will be censored at the last evaluable assessment date.
Overall Survival (OS) | Up to 102 weeks
  The Overall Survival (OS) is defined as the time from first dosing (C1D1) to date of death from any cause. Patients who have not died while on study will be censored at the last evaluable assessment date

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, MD, Principal Investigator — Universitätsklinikum Essen
Locations (7):
- Germany (6):
  - Universitätsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum der Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Istituto Nazionale Tumori Fondazione "G. Pascale", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No